CLINICAL TRIAL: NCT01828970
Title: Glycemic Control Assessed by Continuous Glucose Monitoring in Hemodialyzed Patients With Diabetes Mellitus Treated Via the Basal-Bolus Detemir-Aspart Insulin Regimen: A Pilot Study
Brief Title: Pilot Study of Glycemic Control in Diabetic Hemodialyzed Patients
Acronym: GlyCEDIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Europeen d'Etude du Diabete (Other)
Collaborators: Novo Nordisk A/S (Industry); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/43
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Hemodialysis; Continuous glucose monitoring; Insulin analogues
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Basal-bolus specific insulin regimen (Experimental): Basal-bolus detemir-aspart insulin regimen in hemodialyzed diabetic patients
  Interventions: Drug: Basal-bolus detemir-aspart insulin regimen

INTERVENTIONS:
Drug: Basal-bolus detemir-aspart insulin regimen — After the first CGM was completed during the conventional anti-diabetic treatment, patients received a rapid-acting insulin analogue before each meal (i.e., aspart) and a basal long-acting insulin analogue (i.e., detemir) once or twice daily. The analogues were titrated for optimal glycemic control. After one month of the aspart and detemir regimen, a physician adapted the insulin doses according to the glucose values observed from the second CGM.
  Other Names: Levemir; Novorapid

SUMMARY:
The purpose of the study is to evaluate the effect of the basal-bolus detemir-aspart insulin regimen coupled with continuous glucose monitoring (CGM) on glycemic control in hemodialyzed patients with diabetes

DETAILED DESCRIPTION:
We conducted a pilot prospective multicenter study in five French centers (Strasbourg University Hospital, Strasbourg Sainte Anne Hospital, Colmar, Mulhouse, Valenciennes) designed to evaluate the feasibility and effects of a 3 month treatment regimen with rapid-acting insulin and basal long-acting insulin analogues (i.e., aspart and detemir, respectively) along with CGM on glucose level control in diabetic hemodialyzed patients.

All patients who were admitted to the nephrology departments and matched the inclusion criteria between January 1st, 2010, and June 30th, 2012, were consecutively included in the study. CGM was used to analyze blood glucose excursions at baseline and 1 and 3 months of treatment. It was started during the first dialysis session and then continued for the next two days at home under ambulatory conditions. The CGM was continued during the next dialysis session. Therefore, in total, CGM (Navigator®; Abbott, Rungis, France) was performed for 54 hours, including two consecutive hemodialysis sessions and at 0, 1, and 3 months of treatment. The probe for the system was subcutaneously inserted at the beginning of the first dialysis session to analyze interstitial glucose, and it was removed at the end of the second dialysis session. Due to the time required for CGM calibration, plasma glucose levels were only partially recorded during the first dialysis session.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 83 years
* diagnosis of type 1 or type 2 diabetes
* treatment with insulin injections or oral hypoglycemic agents
* HbA1c ≥ 7% (i.e., 53 mmol/mol)
* on hemodialysis for more than three months

Exclusion Criteria:

* unstable anemia or blood transfusions within the two months prior to the beginning of the study
* a life expectancy of less than 1 year
* chronic inflammatory disease
* evolutive cancer requiring steroid treatment, chemotherapy, radiotherapy, or programmed surgery
* noncompliant patients

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Mean plasma glucose level measured 3 times just before the first hemodialysis session | Baseline and at 3 months of treatment
  Determination by the glucose dehydrogenase method

SECONDARY OUTCOMES:
HbA1c | Baseline and at 3 months of treatment
  Measured by high-performance liquid chromatography
Body weight | Baseline and at 1 month and 3 months of treatment
Insulin requirements | Baseline and at 1 month and 3 months of treatment
  IU per day
Symptomatic hypoglycemia | Baseline and at 1 month and 3 months of treatment
  Number of glycemia < 60 mg/dl per patient and per month
Continuous glucose monitoring parameters | Baseline and at 1 month and 3 months of treatment
  Including: mean continuous glucose monitoring glucose values, within-subjects standard deviation (wSD) and coefficient of variation (wCV = wSD/mean), mean amplitude of glycemic excursion (MAGE), frequency of glucose values under 60 mg/dl, and frequency of glucose values higher than 180 mg/dl
Deaths and major cardiovascular events | Baseline and at 3 months of treatment
  All-cause mortality Major cardiovascular events including: myocardial infarction, stroke, and peripheral vascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Kessler, PhD, Study Director — University Hospital of Strasbourg
Locations (5):
- France (5):
  - Regional Hospital of Colmar, Colmar
  - Regional Hospital of Mulhouse, Mulhouse
  - Sainte Anne Hospital, Strasbourg
  - University Hospital of Strasbourg, Strasbourg
  - Regional Hospital of Valenciennes, Valenciennes

REFERENCES:
- [Background] U S Renal Data System, USRDS 2012 Annual Data Report: Atlas of Chronic Kidney Disease and End-Stage Renal Disease in the United States, National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD, 2012. Available from http://www.usrds.org/atlas.aspx
- [Background] Heras M, Fernandez-Reyes MJ, Sanchez R, Guerrero MT, Molina A, Rodriguez MA, Alvarez-Ude F. Elderly patients with chronic kidney disease: outcomes after 5 years of follow-up. Nefrologia. 2012 May 14;32(3):300-5. doi: 10.3265/Nefrologia.pre2012.Jan.10994. Epub 2012 Feb 28. English, Spanish. PMID 22508140
- [Background] Pieringer H, Biesenbach G. Hemodialysis in patients older than 65 years with end-stage renal failure--comparison of outcome in patients with and without diabetes. Z Gerontol Geriatr. 2008 Apr;41(2):139-45. doi: 10.1007/s00391-007-0467-x. Epub 2008 Mar 11. PMID 18327697
- [Background] Sattar A, Argyropoulos C, Weissfeld L, Younas N, Fried L, Kellum JA, Unruh M. All-cause and cause-specific mortality associated with diabetes in prevalent hemodialysis patients. BMC Nephrol. 2012 Oct 1;13:130. doi: 10.1186/1471-2369-13-130. PMID 23025844
- [Background] Oomichi T, Emoto M, Tabata T, Morioka T, Tsujimoto Y, Tahara H, Shoji T, Nishizawa Y. Impact of glycemic control on survival of diabetic patients on chronic regular hemodialysis: a 7-year observational study. Diabetes Care. 2006 Jul;29(7):1496-500. doi: 10.2337/dc05-1887. PMID 16801568
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] McMurray SD, Johnson G, Davis S, McDougall K. Diabetes education and care management significantly improve patient outcomes in the dialysis unit. Am J Kidney Dis. 2002 Sep;40(3):566-75. doi: 10.1053/ajkd.2002.34915. PMID 12200809
- [Background] Okada T, Nakao T, Matsumoto H, Shino T, Nagaoka Y, Tomaru R, Wada T. Association between markers of glycemic control, cardiovascular complications and survival in type 2 diabetic patients with end-stage renal disease. Intern Med. 2007;46(12):807-14. doi: 10.2169/internalmedicine.46.6355. Epub 2007 Jun 15. PMID 17575371
- [Background] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Background] ACCORD Study Group; Cushman WC, Evans GW, Byington RP, Goff DC Jr, Grimm RH Jr, Cutler JA, Simons-Morton DG, Basile JN, Corson MA, Probstfield JL, Katz L, Peterson KA, Friedewald WT, Buse JB, Bigger JT, Gerstein HC, Ismail-Beigi F. Effects of intensive blood-pressure control in type 2 diabetes mellitus. N Engl J Med. 2010 Apr 29;362(17):1575-85. doi: 10.1056/NEJMoa1001286. Epub 2010 Mar 14. PMID 20228401
- [Background] Riveline JP, Teynie J, Belmouaz S, Franc S, Dardari D, Bauwens M, Caudwell V, Ragot S, Bridoux F, Charpentier G, Marechaud R, Hadjadj S. Glycaemic control in type 2 diabetic patients on chronic haemodialysis: use of a continuous glucose monitoring system. Nephrol Dial Transplant. 2009 Sep;24(9):2866-71. doi: 10.1093/ndt/gfp181. Epub 2009 Apr 23. PMID 19389864
- [Background] Kazempour-Ardebili S, Lecamwasam VL, Dassanyake T, Frankel AH, Tam FW, Dornhorst A, Frost G, Turner JJ. Assessing glycemic control in maintenance hemodialysis patients with type 2 diabetes. Diabetes Care. 2009 Jul;32(7):1137-42. doi: 10.2337/dc08-1688. Epub 2009 Feb 5. PMID 19196889
- [Background] Vos FE, Schollum JB, Coulter CV, Manning PJ, Duffull SB, Walker RJ. Assessment of markers of glycaemic control in diabetic patients with chronic kidney disease using continuous glucose monitoring. Nephrology (Carlton). 2012 Feb;17(2):182-8. doi: 10.1111/j.1440-1797.2011.01517.x. PMID 21883672
- [Background] Ersoy A, Ersoy C, Altinay T. Insulin analogue usage in a haemodialysis patient with type 2 diabetes mellitus. Nephrol Dial Transplant. 2006 Feb;21(2):553-4. doi: 10.1093/ndt/gfi205. Epub 2005 Oct 12. No abstract available. PMID 16221693
- [Background] Schmitz O, Alberti KG, Orskov H. Insulin resistance in uraemic insulin-dependent diabetics. Effect of dialysis therapy as assessed by the artificial endocrine pancreas. Acta Endocrinol (Copenh). 1984 Mar;105(3):371-8. doi: 10.1530/acta.0.1050371. PMID 6367331
- [Background] Simic-Ogrizovic S, Backus G, Mayer A, Vienken J, Djukanovic L, Kleophas W. The influence of different glucose concentrations in haemodialysis solutions on metabolism and blood pressure stability in diabetic patients. Int J Artif Organs. 2001 Dec;24(12):863-9. PMID 11831591
- [Background] Biesenbach G, Raml A, Schmekal B, Eichbauer-Sturm G. Decreased insulin requirement in relation to GFR in nephropathic Type 1 and insulin-treated Type 2 diabetic patients. Diabet Med. 2003 Aug;20(8):642-5. doi: 10.1046/j.1464-5491.2003.01025.x. PMID 12873291
- [Background] Cano N. Bench-to-bedside review: glucose production from the kidney. Crit Care. 2002 Aug;6(4):317-21. doi: 10.1186/cc1517. Epub 2002 Jun 7. PMID 12225606
- [Background] Cersosimo E, Garlick P, Ferretti J. Renal substrate metabolism and gluconeogenesis during hypoglycemia in humans. Diabetes. 2000 Jul;49(7):1186-93. doi: 10.2337/diabetes.49.7.1186. PMID 10909977
- [Background] Abe M, Kaizu K, Matsumoto K. Evaluation of the hemodialysis-induced changes in plasma glucose and insulin concentrations in diabetic patients: comparison between the hemodialysis and non-hemodialysis days. Ther Apher Dial. 2007 Aug;11(4):288-95. doi: 10.1111/j.1744-9987.2007.00492.x. PMID 17661835
- [Background] Chujo K, Shima K, Tada H, Oohashi T, Minakuchi J, Kawashima S. Indicators for blood glucose control in diabetics with end-stage chronic renal disease: GHb vs. glycated albumin (GA). J Med Invest. 2006 Aug;53(3-4):223-8. doi: 10.2152/jmi.53.223. PMID 16953058
- [Background] Holmes G, Galitz L, Hu P, Lyness W. Pharmacokinetics of insulin aspart in obesity, renal impairment, or hepatic impairment. Br J Clin Pharmacol. 2005 Nov;60(5):469-76. doi: 10.1111/j.1365-2125.2005.02476.x. PMID 16236036
- [Background] Rave K, Heise T, Pfutzner A, Heinemann L, Sawicki PT. Impact of diabetic nephropathy on pharmacodynamic and Pharmacokinetic properties of insulin in type 1 diabetic patients. Diabetes Care. 2001 May;24(5):886-90. doi: 10.2337/diacare.24.5.886. PMID 11347749
- [Background] Morello CM. Pharmacokinetics and pharmacodynamics of insulin analogs in special populations with type 2 diabetes mellitus. Int J Gen Med. 2011;4:827-35. doi: 10.2147/IJGM.S26889. Epub 2011 Dec 12. PMID 22267935
- [Background] Meneghini LF, Rosenberg KH, Koenen C, Merilainen MJ, Luddeke HJ. Insulin detemir improves glycaemic control with less hypoglycaemia and no weight gain in patients with type 2 diabetes who were insulin naive or treated with NPH or insulin glargine: clinical practice experience from a German subgroup of the PREDICTIVE study. Diabetes Obes Metab. 2007 May;9(3):418-27. doi: 10.1111/j.1463-1326.2006.00674.x. PMID 17391170
- [Background] Marshall J, Jennings P, Scott A, Fluck RJ, McIntyre CW. Glycemic control in diabetic CAPD patients assessed by continuous glucose monitoring system (CGMS). Kidney Int. 2003 Oct;64(4):1480-6. doi: 10.1046/j.1523-1755.2003.00209.x. PMID 12969169
- [Background] Tzamaloukas AH, Yuan ZY, Murata GH, Balaskas E, Avasthi PS, Oreopoulos DG. Clinical associations of glycemic control in diabetics on CAPD. Adv Perit Dial. 1993;9:291-4. PMID 8105946
- [Result] Shurraw S, Hemmelgarn B, Lin M, Majumdar SR, Klarenbach S, Manns B, Bello A, James M, Turin TC, Tonelli M; Alberta Kidney Disease Network. Association between glycemic control and adverse outcomes in people with diabetes mellitus and chronic kidney disease: a population-based cohort study. Arch Intern Med. 2011 Nov 28;171(21):1920-7. doi: 10.1001/archinternmed.2011.537. PMID 22123800
- [Result] Hendriksen KV, Jensen T, Oturai P, Feldt-Rasmussen B. Effects of insulin detemir and NPH insulin on renal handling of sodium, fluid retention and weight in type 2 diabetic patients. Diabetologia. 2012 Jan;55(1):46-50. doi: 10.1007/s00125-011-2345-8. Epub 2011 Oct 16. PMID 22002075